CLINICAL TRIAL: NCT03992365
Title: A Prospective, Randomized, Evaluator Blind, Active-Controlled, Parallel Study of the Efficacy and Safety of Quiklean® and Klean-Prep With Dulcolax® for the Bowel Preparation Prior to Colonoscopy
Brief Title: Study of the Efficacy and Safety of Quiklean® and Klean-Prep With Dulcolax® for the Bowel Preparation Prior to Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universal Integrated Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UIC-STP-2017
Record Dates: First submitted 2019-06-06; First posted 2019-06-20 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Bowel Preparation
Keywords: non-inferiority
MeSH Terms: interventions — sodium phosphate; polyethylene glycol 3350; Sodium Bicarbonate; Sodium Chloride; Potassium Chloride

STUDY DESIGN:
Intervention Model Description: randomized, evaluator blind, active-controlled, parallel study
Who Masked: Outcomes Assessor
Masking Description: After bowel preparation, independent evaluator who is blinded to subject's treatment will evaluate the overall colon cleansing based on Aronchick and Ottawa scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quiklean® (Experimental): Quiklean® (32 tablets)
  Interventions: Drug: Quiklean® (sodium phosphate monobasic monohydrate, USP, and sodium phosphate dibasic anhydrous, USP)
- GroKlean-Prep with Dulcolax® (Active Comparator): 2 sachets of Klean-Prep with 1 tablet of Dulcolax®
  Interventions: Drug: Polyethylene glycol 3350, sodium sulfate anhydrous, sodium bicarbonate, sodium chloride, potassium chloride, aspartame;Bisacodyl

INTERVENTIONS:
Drug: Quiklean® (sodium phosphate monobasic monohydrate, USP, and sodium phosphate dibasic anhydrous, USP) — The evening before the colonoscopy: Take 4 tablets with 250 ml of clear liquids every 15 minutes for a total of 20 tablets.
  On the day of the colonoscopy: Starting 3-5 hours before the procedure, take 4 tablets with 250 ml of clear liquids every 15 minutes for a total of 12 tablets.
  Other Names: sodium phosphate
  Arms: Quiklean®
Drug: Polyethylene glycol 3350, sodium sulfate anhydrous, sodium bicarbonate, sodium chloride, potassium chloride, aspartame;Bisacodyl — The day before the colonoscopy: One 5 mg tablet of Dulcolax® will be administered, do not chew or crush the tablet, in the afternoon before the day of colonoscopy. About 4 hours after administration of Dulcolax®, drink the 1000 ml Klean-Prep solution at a rate of 250 ml every 15 minutes.
  On the day of the colonoscopy: Starting 3-5 hours before the procedure, drink the 1000 ml Klean-Prep solution at a rate of 250 ml every 15 minutes.
  Other Names: PEG
  Arms: GroKlean-Prep with Dulcolax®

SUMMARY:
The objective is to demonstrate that investigational drug, Quiklean®, is not inferior to standard comparator, Klean-Prep with Dulcolax®, with respect to the overall quality of bowel preparation in subjects undergoing colonoscopy.

DETAILED DESCRIPTION:
This will be a randomized, evaluator blind, active-controlled, parallel study to compare the safety and efficacy of investigational drug (Quiklean®) with standard comparator (Klean-Prep with Dulcolax®) in subjects undergoing bowel preparation for colonoscopy. This study will be conducted in two arms:

1. Group A: Quiklean® (32 tablets)
2. Group B: 2 sachets of Klean-Prep with 1 tablet of Dulcolax® The study will be consist of 4 clinical visits. Subjects will come to the clinics at Visit 1 (the start of the screening), Visit 2 (randomization), and Visit 3 (colonoscopy visit), and Visit 4 (follow-up visit) according to the pre-defined schedule.

After the inform consent is obtained from the subject, the designated assessment will be performed. If the eligibility criteria has been met, the subjects will be randomly assigned with a 1:1 (Group A:B) and scheduled to a colonoscopy. The colonoscopy visit should be arranged within 10 days after screening visit and randomization. Subjects are instructed how to take study medication, and standard dietary instructions for each group are identical.

After bowel preparation, the colonoscopy will be performed in the morning by the experienced colonoscopist, and the entire process of colonoscopy will be simultaneously recorded by video. The quality of bowel cleansing in video will be rated by an independent blinded colonoscopist after the completion of colonoscopy.

The modified Aronchick scale for the primary efficacy endpoint and the Ottawa scale, and subject's responses to the acceptability and tolerability for the secondary efficacy endpoint will be rated and collected. The safety laboratory examinations from the blood sample, solicited events from the start of administration of study medications before colonoscopy, and treatment-emergent adverse events will be also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 20 and 74 years of age.
2. Subject who are scheduled for an elective colonoscopy.
3. Ability to complete the entire procedure and to comply with study instructions.
4. Will provide completed and signed written informed consents.

Exclusion Criteria:

1. Subjects with severe chronic constipation, defined as fewer than one bowel movement per week for a period > 1 year.
2. Subjects with known or suspected acute exacerbation of chronic inflammatory bowel disease (IBD).
3. Subjects with significant gastrointestinal disease, such as gastrointestinal obstruction or perforation, active ulcerative colitis, toxic colitis, and toxic megacolon.
4. Subjects with ascites of any etiology.
5. Subjects with renal insufficiency, defined as serum creatinine > 1.5 times the upper limit of normal (ULN).
6. Subjects with current or history of abdominal surgeries as follow:

   * Acute surgical abdominal conditions.
   * Any prior colorectal surgery within previous 3 months at screening, excluding appendectomy, hemorrhoid surgery or prior endoscopic procedures.
   * History of ileostomy, right or transverse colostomy, subtotal colectomy with ileosimoidostomy, with ≥ 50% of colon removed, excluding right or left hemicolectomy.
   * History of gastric bypass or stapling history.
7. Subjects with any serious cardiovascular diseases or related interventions as follows:

   * History or current evidence of prolonged QT, unstable angina pectoris, untreated arrhythmia, or uncontrolled hypertension, cardiomyopathy, congestive heart failure (New York Heart Association (NYHA) Functional Classification, grades 3 and 4).
   * Myocardial Infarction (MI) within previous 3 months at screening.
   * Percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass graft surgery within previous 3 months at screening.
   * Subject has undergone cardiovascular stent procedure or carotid artery stenting procedure, and continues to receive an anticoagulant regimen within 1 year prior to screening.
   * Current use digitalis preparations or any medications known to prolong QT interval.
8. Subjects with history of seizures or at risk of seizure, such as subjects taking medications that lower the seizure threshold (e.g., tricyclic antidepressants), or subjects withdrawing from alcohol or benzodiazepines, subjects with known or suspected hyponatremia.
9. Subject has clinically significant abnormal laboratory values of electrolytes at screening, including phosphorus, sodium, potassium, calcium, chloride, and magnesium.
10. Subjects with history of biopsy-proven acute phosphate nephropathy.
11. Subjects with history of phenylketonuria.
12. Subject has severe dehydration, or severe abdominal pain associated with nausea and vomiting at screening.
13. Subject has problems with swallowing or gastric reflux, or subjects is at risk of aspiration.
14. Subjects is pregnant, lactating women or women of childbearing potential without an effective method of birth control (e.g. oral contraceptive, intrauterine device, surgical sterilization, hysterectomy).
15. Subjects with hypersensitivity to any ingredients in the study medications.
16. Participation in any other investigational study within 30 days prior to receiving study medication.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Aronchick scale | up to 24 weeks
  The percentage of subjects that achieve excellent or good cleansing (success rate) in the Aronchick Scale.

SECONDARY OUTCOMES:
Ottawa scale | up to 24 weeks
  Proportion of successes (excellent, good, or fair) by individual colon segment (ascending, transverse, descending), which are assessed with the Ottawa scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Liang Chen, Dr, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No